CLINICAL TRIAL: NCT05005988
Title: Actions for Empowered Maternal Neonatal Care (ACUNE): Nursing Intervention to Strengthen Mothers' Competence to Care for Their Preterm Infants at Home. A Pilot Study
Brief Title: Actions for Empowered Maternal Neonatal Care (ACUNE): A Nursing Intervention
Acronym: ACUNE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, SANDRA PATRICIA OSORIO GALEANO, Principal Investigator, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEI-FE2020-02
Record Dates: First submitted 2021-08-02; First posted 2021-08-16 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-08

CONDITIONS: Patient Empowerment
Keywords: Health education; Discharge patient; Neonatal Nursing; Neonatal Intensive Care Unit
MeSH Terms: conditions — Patient Participation; Health Education

STUDY DESIGN:
Intervention Model Description: Single-blinded, parallel, randomized clinical trial. Mothers in the intervention group will receive a pre-discharge empowerment educational intervention, and the control group will receive the usual discharge preparation. Three 30-minute sessions will be conducted with each mother in the intervention group, the first during the first week after admission, the second session within 7 days after the second session, and the third 3 to 2 days before discharge. An induction to the out-of-hospital kangaroo program will also take place on the day of admission to the program. Mothers will receive a booklet with general care contents and empowerment information. Mothers in the control group will receive the usual preparation for discharge from the NICU. Response variables will be measured at three time points: At admission (baseline), before discharge and one week after the discharge.
Who Masked: Outcomes Assessor
Masking Description: The outcome evaluator will be external to the intervention and will not know whether the mothers belong to the intervention or control group. This person will be trained and standardized in the handling of the instruments, will know the general elements of the study, and will ensure compliance with the ethical conditions established in the study.
  Outcome evaluator will be informed at the time of applying the instruments and recording the information related to the variables of interest of the study and will verify the complete filling out of the instruments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empowerment educational intervention (Experimental): Three 30-minute sessions will be conducted with each mother in the intervention group, the first during the first week after admission, the second session within 7 days after the second session, and the third 3 to 2 days before discharge. An induction to the out-of-hospital kangaroo program will also take place on the day of admission to the program. Mothers will receive a booklet with general care contents and empowerment information.
  Interventions: Behavioral: Actions for Empowered Maternal Neonatal Care
- Usual intervention (No Intervention): Mothers receive information for home infant care, no theoretical perspective and no empowerment approach is considered

INTERVENTIONS:
Behavioral: Actions for Empowered Maternal Neonatal Care — The intervention includes three 30-minute face-to-face sessions:
  Session 1. Recognizing prematurity and the NICU environment: includes definitions of prematurity, characteristics of premature infants, equipment and dynamics of NICU care. Mothers are encouraged to identify their own and contextual resources that can help empower them.
  Session 2. Identifying the care of a premature baby: aspects related to the kangaroo method, feeding, thermoregulation, among others, are presented. Knowledge is presented as an empowerment resource.
  Session 3: Preparation for the return home. Aspects related to the discharge process and transition to home are described. Includes information on the transition home, warning signs, emergency situations, physical burden, and recognition of sources of personal and professional support.
  Session on admission to the out-of-hospital kangaroo program: presents the dynamics of the kangaroo program, as well as the goals in the new care setting.
  Other Names: ACUNE
  Arms: Empowerment educational intervention

SUMMARY:
The quality of care premature infants receive at home after hospital discharge is critical to their health and well-being. Premature infants require special care, which is why Neonatal Intensive Care Units (NICUs) have processes in place to prepare mothers for discharge. However, this experience is very complex for mothers, who often experience high levels of stress, anxiety, sadness and uncertainty. Mothers need knowledge and skills about caring for a premature infant, but they also need to gain confidence, believe in their abilities, and become empowered to participate more actively and confidently in decisions that have to do with their child's health. Several approaches exist to prepare mothers for home-based infant care; in the present study, an intervention focused on empowerment is proposed as a way to strengthen mothers' competence to care for their preterm infants and improve infant health outcomes. The intervention is expected to have adequate acceptability and feasibility, as well as preliminary evidence that it improves mothers' competence to care for their infants and decreases readmissions, emergency department visits, improves weight gain and health outcomes of preterm infants.

DETAILED DESCRIPTION:
Premature children have a higher risk of becoming ill and dying than full-term children and that risk do not end with hospitalization, so the care they receive at home is decisive in their health and wellbeing. Preterm infants are especially vulnerable and have a greater number of readmissions and emergency visits after discharge, as well as delays in vaccination, infections as well as nutritional alterations.

Women play central in family health, and it is necessary to design and applying interventions to facilitate a woman's empowerment, specially to care premature son at home after Neonatal Intensive Care Units (NICU) discharge. Preparation for discharge has been described in the literature as a process where the mothers develop skills and knowledge that they will need to care for their premature children once they are at home. However, for mothers, they face a challenging task in which they experience high levels of stress, fear and uncertainty. Premature children require particular care and the mothers need more than knowledge and skills, they also need to get confidence, believe in their abilities and empowerment themselves to participate more actively and safely in decisions that have to do with the health of their children. This study arises from the need to prepare mothers through the possibilities of empowerment, as a way to improve the health outcomes of premature children. A Randomized Clinical Trial is proposed to establish the effect of the educational intervention of empowerment on mothers' competence in premature infant care, readmissions, weight gain, exclusive breastfeeding and other aspects related to the health, survival and well-being of premature infants. The intervention was designed by integrating the theoretical approach, empirical evidence and the results of a qualitative study in which mothers and fathers of premature infants participated, which gives a participatory approach to the research and makes it close to the parents' reality and gives it social relevance.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of premature infants less than 37 weeks gestational age at birth.
* Mothers of premature infants hospitalized in the neonatal intensive care unit

Exclusion Criteria:

* Mothers with previous experience in caring for a premature infant.
* Mothers whose children have some type of congenital malformation.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in the caregiver's competence | At admission (baseline), through hospitalization completion, an average of 3 week and one week after the discharge.
  The caregiver's competence is the capacity, ability and preparation that the caregiver has to perform his or her caregiving task at home and can be measured with the CUIDAR scale, which was designed and validated in Colombia. This scale has been used in several studies, confirming its validity and reliability. To determine the validity and reliability of the CUIDAR instrument in mothers of premature infants, a cross-sectional quantitative study was carried out in which its psychometric properties were measured. 207 mothers of premature infants participated. A factor analysis did not confirm the original structure in the new population, but a model with 7 factors and 33 items with a Cronbach's alpha of 0.852 and adequate goodness-of-fit indices. The new version of the scale, named CUIDAR-PreMa, has 7 dimensions: Acting, Coping, Bonding, Social Support, General Knowledge, Singularity and Specific Knowledge. The scale has 33 items, with a Likert-type scale

SECONDARY OUTCOMES:
Change in premature infant body weight | At admission (baseline), through hospitalization completion, an average of 3 week and one week after the discharge.
  Weight of the premature infant in grams. Measurements obtained by the percentile curve are evaluated.
Readmission | One week after the discharge
  Readmission iin the week following hospital discharge
Emergency visits | One week after discharge
  Emergency visits number in the firts week after discharge
Exclusive breastfeeding | One week after discharge
  Exclusive breastfeeding refers to whether the mother covers all of her child's feeding needs with breast milk. To establish this, a questionnaire will be used to determine how many times a day she expresses breast milk and how many cubic centimeters of breast milk she expresses, whether the premature child has a good suckling ability and whether she has had to give her child formula milk to supplement his or her diet.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra P Osorio Galeano, MD, Principal Investigator — Universidad de Antioquia; Angela M Salazar Maya, PhD, Study Director — Universidad de Antioquia
Locations (1):
- Sandra Osorio, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osorio Galeano SP, Salazar Maya AM. Experiences of Parents of Preterm Children Hospitalized Regarding Restrictions to Interact with Their Children Imposed Because of the COVID-19 Pandemic. Invest Educ Enferm. 2021 Jun;39(2):e10. doi: 10.17533/udea.iee.v39n2e10. PMID 34214287
- [Derived] Osorio-Galeano SP, Salazar-Maya AM. Design and assessment of an intervention for parents of premature newborns: a mixed-methods study. Rev Lat Am Enfermagem. 2026 Feb 2;34:e4747. doi: 10.1590/1518-8345.7791.4747. eCollection 2026. PMID 41637376